CLINICAL TRIAL: NCT00009698
Title: IL-2 Infusion in AML Patients After Autologous Bone Marrow Transplant: A Pediatric Oncology Group Wide Phase I Trial
Brief Title: Interleukin-2 in Treating Children Who Have Undergone Bone Marrow Transplantation for Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9674; POG-9674 (Other: Pediatric Oncology Group); CDR0000065574 (Other: Clinical Trials.gov)
Record Dates: First submitted 2001-02-02; First posted 2003-12-31 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2)
MeSH Terms: conditions — Leukemia | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Day 1 through day 7, days 9-14 and days 16-22: The assigned dose of IL-2 will be administered SQ. On days 8 and 15, IL-2 will be administered as a 2 hour intravenous infusion of one million units/M2 of IL-2. After day 22 there will be a 7 day rest period before beginning the next cycle. The next cycle will repeat just as above. This will be repeated for a maximum of 4 total cycles of 21 days of IL-2 therapy. The maintenance dose of IL-2 will always be the same as given during cycle one, unless there is dose limiting toxicity.
  Interventions: Biological: aldesleukin

INTERVENTIONS:
Biological: aldesleukin — Given SQ and IV
  Other Names: Recombinant Interleukin-2 (Chiron-Cetus) (IL-2); NSC -373364

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-2 in treating children who have undergone bone marrow transplantation for acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of interleukin-2 after autologous bone marrow transplantation in pediatric patients with acute myeloid leukemia. II. Determine toxic effects of this regimen in these patients.

OUTLINE: This is a dose escalation study. Patients receive interleukin-2 (IL-2) subcutaneously on days 1-7, 9-14, and 16-22. On days 8 and 15, patients receive IL-2 IV over 2 hours. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 6-9 patients receive escalating doses of IL-2 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 2 of 9 patients experience dose-limiting toxicity. Patients are followed every 6 months for 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of acute myeloid leukemia (AML) Must have received autologous bone marrow or stem cell transplantation for AML within the past 28 to 100 days Evidence of marrow engraftment Absolute neutrophil count at least 500/mm3 for at least 2 consecutive days Platelet count at least 20,000/mm3 without transfusion support for more than 3 days Documented M1 or M2 bone marrow within the past 7 days

PATIENT CHARACTERISTICS: Age: Under 22 at diagnosis Performance status: Karnofsky 50-100% Life expectancy: At least 8 weeks Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 1.5 mg/dL SGPT no greater than 2 times normal Renal: Creatinine normal OR Glomerular filtration rate at least 70 mL/min Cardiovascular: Shortening fraction at least 27% OR Ejection fraction greater than 50% No evidence of active cardiac disease by electrocardiogram Pulmonary: No evidence of active pulmonary disease by chest x-ray Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Neurologic deficits due to CNS disease must be stable within the past 4 weeks No active viral, bacterial, or invasive fungal infection No fever No prior hypersensitivity to interleukin-2 No greater than grade 2 mucosal toxicity

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 3 days since prior growth factors or intravenous immunoglobulin No concurrent cytokines or growth factors No concurrent intravenous immunoglobulin Chemotherapy: No concurrent chemotherapy No concurrent methotrexate IV or intrathecally Endocrine therapy: At least 3 days since prior corticosteroids No concurrent corticosteroids (except as premedication for documented severe transfusion reactions) Radiotherapy: Not specified Surgery: Not specified Other: At least 3 days since prior pentoxifylline or amphotericin B No concurrent pentoxifylline No other concurrent anticancer therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 1998-03; Primary Completion 2001-06 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of IL-2 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kimo C. Stine, MD, Study Chair — Arkansas Children's Hospital at the University of Arkansas for Medical Sciences
Locations (119):
- United States (104):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - University of Miami-Jackson Memorial Hospital Medical Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - CCOP - Florida Pediatric, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Texas Oncology P.A., Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - MBCCOP - South Texas Pediatric, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School-Charleston, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Clinique de Pediatrie, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne